CLINICAL TRIAL: NCT01712516
Title: A 12-week Treatment, Multi-center, Randomized, Double-blind, Parallel-group, Placebo and Active Controlled Study to Assess the Efficacy, Safety, and Tolerability of Indacaterol Maleate / Glycopyrronium Bromide in COPD Patients With Moderate to Severe Airflow Limitation
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CQVA149A2337
Record Dates: First submitted 2012-10-19; First posted 2012-10-23 (Estimated); Results first posted 2015-07-15 (Estimated); Last update posted 2015-07-15 (Estimated); Status verified 2015-07

CONDITIONS: Chronic Obstructive Pulmonary Disease (COPD)
Keywords: COPD, QVA149
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — indacaterol-glycopyrronium combination; indacaterol; Glycopyrrolate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- QVA149 (Experimental): 27.5/12.5 ug twice daily (b.i.d.) Single Dose Dry Powder Inhaler (SDDPI
  Interventions: Drug: QVA149
- QAB149 (Active Comparator): 27.5 ug b.i.d.
  Interventions: Drug: QAB149
- NVA237 (Active Comparator): 12.5 ug b.i.d.
  Interventions: Drug: NVA237
- Placebo (Placebo Comparator): b.i.d.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: QVA149 — QVA149 was supplied in a capsule form in blister packs for use in the Novartis Concept1 SDDPI
  Arms: QVA149
Drug: QAB149 — QAB149 was supplied in capsule form in blister packs for use in the Novartis Concept1 SDDPI.
  Arms: QAB149
Drug: NVA237 — NVA237 was supplied in capsule form in blister packs for use in the Novartis Concept1 SDDPI.
  Arms: NVA237
Drug: Placebo — Placebo was supplied in capsule form in blister packs for use in the Novartis Concept1 SDDPI.
  Arms: Placebo

SUMMARY:
This study will assess the efficacy, safety and tolerability of indacaterol maleate/glycopyrronium bromide in patients with moderate to severe airflow limitation.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients that have signed informed consent and are >/= 40 years of age.
* Patients with stable COPD according to GOLD 2011.
* Patients with a post-bronchodilator FEV1 of >/= 30% and < 80% predicted and a post-bronchodilator FEV1/FVC <0.70.
* Current or ex-smokers who have a smoking history of at least 10 pack years.
* Patients with an mMRC grade 2 or greater.

Exclusion Criteria:

* Patients with Type I or uncontrolled Type II diabetes - Patients with a history of long QT syndrome or whose QTc measured at Visit 101 (Fridericia method) is prolonged (>450 ms for males and females) and confirmed by a central assessor. (These patients should not be re-screened.)
* Patients who have a clinically significant ECG abnormality at Visit 101 or Visit 102. (These patients should not be re-screened.)
* Patients with a history of malignancy of any organ system, treated or untreated, within the last five years.
* Patients with narrow-angle glaucoma, BPH or bladder-neck obstruction or moderate-severe renal impairment or urinary retention.
* Patients who had a COPD exacerbation within 6 weeks prior to screening.
* Patients who have a respiratory tract infection within 4 weeks prior to screening.
* Patients requiring long term oxygen therapy prescribed for more than 12 hr per day.
* Patients with a history of asthma. 8. Patients with an onset of respiratory symptoms, including COPD diagnosis, prior to age 40 years.
* Patients with a blood eosinophil count of greater than 600 mm/3 during run-in.
* Patients with concomitant pulmonary disease.
* Patients with a diagnosis of alpha-1 anti-trypsin deficiency.
* Patients with active pulmonary tuberculosis.
* Patients in the active phase of a pulmonary rehabilitation programme.
* Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1001 (Actual)
Dates: Start 2012-12; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (85):
- United States (49):
  - Novartis Investigative Site, Huntsville, Alabama
  - Novartis Investigative Site, *See Various Dept.'s*, Arizona
  - Novartis Investigative Site, Tempe, Arizona
  - Novartis Investigative Site, Buena Park, California
  - Novartis Investigative Site, Fullerton, California
  - Novartis Investigative Site, Palmdale, California
  - Novartis Investigative Site, Riverside, California
  - Novartis Investigative Site, San Diego, California
  - Novartis Investigative Site, Sepulveda, California
  - Novartis Investigative Site, Clearwater, Florida
  - Novartis Investigative Site, DeLand, Florida
  - Novartis Investigative Site, Fort Lauderdale, Florida
  - Novartis Investigative Site, Miami, Florida
  - Novartis Investigative Site, Orlando, Florida
  - Novartis Investigative Site, Pensacola, Florida
  - Novartis Investigative Site, Port Orange, Florida
  - Novartis Investigative Site, Sarasota, Florida
  - Novartis Investigative Site, Tamarac, Florida
  - Novartis Investigative Site, Tampa, Florida
  - Novartis Investigative Site, Winter Park, Florida
  - Novartis Investigative Site, Lawrenceville, Georgia
  - Novartis Investigative Site, Opelousas, Louisiana
  - Novartis Investigative Site, Henderson, Nevada
  - Novartis Investigative Site, Las Vegas, Nevada
  - Novartis Investigative Site, Reno, Nevada
  - Novartis Investigative Site, Brandon, New Jersey
  - Novartis Investigative Site, Charlotte, North Carolina
  - Novartis Investigative Site, Huntersville, North Carolina
  - Novartis Investigative Site, Raleigh, North Carolina
  - Novartis Investigative Site, Shelby, North Carolina
  - Novartis Investigative Site, Charleston, South Carolina
  - Novartis Investigative Site, Columbia, South Carolina
  - Novartis Investigative Site, Easley, South Carolina
  - Novartis Investigative Site, Gaffney, South Carolina
  - Novartis Investigative Site, Greenville, South Carolina
  - Novartis Investigative Site, Pelzer, South Carolina
  - Novartis Investigative Site, Rock Hll, South Carolina
  - Novartis Investigative Site, Seneca, South Carolina
  - Novartis Investigative Site, Simpsonville, South Carolina
  - Novartis Investigative Site, Spartanburg, South Carolina
  - Novartis Investigative Site, Union, South Carolina
  - Novartis Investigative Site, Johnson City, Tennessee
  - Novartis Investigative Site, Arlington, Texas
  - Novartis Investigative Site, Corsicana, Texas
  - Novartis Investigative Site, Dallas, Texas
  - Novartis Investigative Site, Fort Worth, Texas
  - Novartis Investigative Site, Lufkin, Texas
  - Novartis Investigative Site, McKinney, Texas
  - Novartis Investigative Site, Tyler, Texas
- Colombia (3):
  - Novartis Investigative Site, Barranquilla, Atlántico
  - Novartis Investigative Site, Armenia
  - Novartis Investigative Site, Barranquilla
- Novartis Investigative Site, Alexandria, Egypt
- France (4):
  - Novartis Investigative Site, Beuvry, France
  - Novartis Investigative Site, Nantes
  - Novartis Investigative Site, Paris
  - Novartis Investigative Site, Reims
- Novartis Investigative Site, Guatemala City, Departamento de Guatemala, Guatemala
- Hungary (11):
  - Novartis Investigative Site, Balassagyarmat, Hungary
  - Novartis Investigative Site, Debrecen, Hungary
  - Novartis Investigative Site, Komárom, Hungary
  - Novartis Investigative Site, Tatabánya, Hungary
  - Novartis Investigative Site, Deszk
  - Novartis Investigative Site, Gödöllő
  - Novartis Investigative Site, Győr
  - Novartis Investigative Site, Makó
  - Novartis Investigative Site, Miskolc
  - Novartis Investigative Site, Százhalombatta
  - Novartis Investigative Site, Szombathely
- Novartis Investigative Site, Panama City, Provincia de Panamá, Panama
- Slovakia (14):
  - Novartis Investigative Site, Bardejov, Slovak Republic
  - Novartis Investigative Site, Bojnice, Slovak Republic
  - Novartis Investigative Site, Humenné, Slovak Republic
  - Novartis Investigative Site, Liptovský Hrádok, Slovak Republic
  - Novartis Investigative Site, Nitra, Slovak Republic
  - Novartis Investigative Site, Vráble, Slovak Republic
  - Novartis Investigative Site, Galanta, Slovakia
  - Novartis Investigative Site, Košice, Slovakia
  - Novartis Investigative Site, Kráľovský Chlmec, Slovakia
  - Novartis Investigative Site, Prešov, Slovakia
  - Novartis Investigative Site, Prievidza, Slovakia
  - Novartis Investigative Site, Zvolen, Slovakia
  - Novartis Investigative Site, Martin
  - Novartis Investigative Site, Spisská Nová Ves
- Novartis Investigative Site, Golnik, Slovenia

REFERENCES:
- [Derived] Mahler DA, Kerwin E, Murray L, Dembek C. The Impact of Twice-Daily Indacaterol/Glycopyrrolate on the Components of Health-Related Quality of Life and Dyspnea in Patients with Moderate-to-Severe Chronic Obstructive Pulmonary Disease. Chronic Obstr Pulm Dis. 2019 Oct 23;6(4):308-20. doi: 10.15326/jcopdf.6.4.2019.0131. PMID 31539467

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were randomized to each treatment arm in a 1:1:1:1 ratio.
Pre-assignment Details: One thousand one participants were randomized. (One participant was randomized twice, took study drug twice and was counted twice in the randomized and safety sets). In the safety set, participants were analyzed according to the treatment received.
Groups:
- QVA149: 27.5/12.5 ug twice daily (b.i.d.) via Single Dose Dry Powder Inhaler (SDDPI)
Period: Overall Study
Arm/Group | QVA149 | QAB149 | NVA237 | Placebo
Started | 250 | 251 | 251 | 249
Safety Set | 250 | 251 | 251 | 248
Full Analysis Set | 250 | 251 | 250 | 247
Completed | 244 | 241 | 245 | 236
Not Completed | 6 | 10 | 6 | 13
Not completed — Technical problems | 0 | 0 | 0 | 2
Not completed — Lost to Follow-up | 0 | 0 | 2 | 1
Not completed — Death | 0 | 1 | 0 | 0
Not completed — Protocol deviation | 1 | 0 | 1 | 0
Not completed — Physician Decision | 2 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 3 | 9 | 3 | 9

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | QVA149 | QAB149 | NVA237 | Placebo | Total
Number analyzed (Participants) | 250 | 251 | 251 | 249 | 1001
Age, Continuous [Mean (Standard Deviation); unit: Years] | 62.8 (8.46) | 63.7 (8.58) | 63.1 (8.53) | 62.5 (8.07) | 63.0 (8.41)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 96 | 101 | 107 | 111 | 415
  Male | 154 | 150 | 144 | 138 | 586

OUTCOME MEASURES:

1. Primary Outcome: Primary: Change From Baseline in Standardized Forced Expiratory Volume in 1 Second (FEV1) Area Under the Curve (AUC) (0-12 Hours (h))
Description: Pulmonary function assessments were performed using centralized spirometry according to international standards. Baseline FEV1 was defined as the average of the pre-dose FEV1 measured at -45 minutes (min) and -15 min at day 1. A mixed model for repeated measures (MMRM), used for this analysis, included terms of treatment, baseline FEV1 measurements, smoking status at baseline, baseline inhaled corticosteroid (ICS) use, region, baseline FEV1 * visit interaction, and visit, treatment * visit interaction. Missing values of FEV1 AUC0-12 at Day 1 and Week 12 will not imputed. The trapezoidal rule was used to calculate FEV1 AUC and then normalized to the length of time.
Time Frame: baseline (BL), 12 weeks
Population: Full Analysis Set: The full analysis set included all randomized participants who received at least one dose of study treatment. Participants, who were missing day 1 and/or week 12 FEV1 AUC 0-12h measurements, were not included in the analysis.
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | QVA149 | QAB149 | NVA237 | Placebo
Number analyzed (Participants) | 249 | 251 | 250 | 246
Liters | 0.234 (0.0134) | 0.122 (0.0134) | 0.155 (0.0134) | -0.028 (0.0137)

2. Secondary Outcome: Change From Baseline in St. George's Respiratory Questionnaire (SGRQ) Total Score
Description: Participants reported change in health status by using the SGRQ. The SGRQ contains 50 items divided into 2 parts covering 3 aspects of health related to COPD: Part I covers "Symptoms" and is concerned with respiratory symptoms, their frequency and severity; Part II covers "Activity" and is concerned with activities that cause or are limited by breathlessness; Part II is also concerned with "Impacts", which covers a range of aspects concerned with social functioning and psychological disturbances resulting from airways disease. A score was calculated for each of these 3 subscales and a "Total" score was calculated. In each case the lowest possible value is zero and the highest 100. Higher values correspond to greater impairment of health status. Missing week 12 data were imputed with Last Observation Carried Forward (LOCF) method but only if measured at day >= 29. A negative change from baseline indicates improvement.
Time Frame: BL, 12 Weeks
Population: Full Analysis Set: The full analysis set included all randomized participants who received at least one dose of study treatment. Participants missing week 12 data were not included in the analysis.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | QVA149 | QAB149 | NVA237 | Placebo
Number analyzed (Participants) | 238 | 234 | 237 | 226
score on a scale | -7.5 (0.85) | -5.9 (0.86) | -6.0 (0.86) | -1.1 (0.88)

3. Secondary Outcome: Percentage of Participants With a Clinically Important Improvement of at Least 4 Units in the SGRQ Total Score
Description: Participants reported change in health status by using the SGRQ. The SGRQ contains 50 items divided into 2 parts covering 3 aspects of health related to COPD: Part I covers "Symptoms" and is concerned with respiratory symptoms, their frequency and severity; Part II covers "Activity" and is concerned with activities that cause or are limited by breathlessness; Part II is also concerned with "Impacts", which covers a range of aspects concerned with social functioning and psychological disturbances resulting from airways disease. A score was calculated for each of these 3 subscales and a "Total" score was calculated. In each case the lowest possible value is zero and the highest 100. Higher values correspond to greater impairment of health status.
Time Frame: 12 weeks
Population: Participants from the full analysis set, who had a SGRQ total score, were included in the analysis. The full analysis set included all randomized participants who received at least one dose of study treatment.
Measure: Number; unit: Percentage of participants
Arm/Group | QVA149 | QAB149 | NVA237 | Placebo
Number analyzed (Participants) | 238 | 234 | 237 | 226
Percentage of participants | 59.2 | 56.8 | 51.5 | 34.5

4. Secondary Outcome: Change From Baseline in Trough FEV1
Description: Pulmonary function assessments were performed using centralized spirometry according to international standards. Trough FEV1 was analyzed using the same MMRM as specified for FEV1. Trough FEV1 was defined as the mean of FEV1 at 23 h 15 min and 23 h 45 min after the morning dose of the previous day. Before the mean was calculated, a time window of 10 - 13 hours post-evening dose was applied to these 2 measurements. Recordings outside the time window were set to missing.
Time Frame: BL, day 2, day 86
Population: Full Analysis Set (FAS): The FAS included all randomized participants who received at least one dose of study treatment. Participants, who had both baseline and post baseline values for a given time point, were included in the analysis for that time point.
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | QVA149 | QAB149 | NVA237 | Placebo
Number analyzed (Participants) | 246 | 251 | 249 | 245
Liters
  day 2 | 0.208 (0.0107) | 0.111 (0.0106) | 0.132 (0.0107) | 0.010 (0.0107)
  day 86 | 0.216 (0.0142) | 0.138 (0.0141) | 0.128 (0.0142) | -0.017 (0.0145)

5. Secondary Outcome: Change From Baseline in Pre-dose Trough FEV1
Description: Pulmonary function assessments were performed using centralized spirometry according to international standards. Pre-dose trough FEV1 was analyzed using the same MMRM as specified for FEV1. Pre-dose trough FEV1 was defined as the mean of FEV1 at -45 min and -15 min before the morning dose. Since the time of evening dose of the previous day was not recorded at these visits, no time window was applied.
Time Frame: BL, day 85
Population: Full Analysis Set (FAS): The FAS included all randomized participants who received at least one dose of study treatment. Participants, who had both baseline and week 12 values, were included in the analysis.
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | QVA149 | QAB149 | NVA237 | Placebo
Number analyzed (Participants) | 243 | 249 | 246 | 241
Liters | 0.193 (0.0132) | 0.100 (0.0132) | 0.108 (0.0133) | -0.027 (0.0135)

6. Secondary Outcome: Change From Baseline in FEV1
Description: Pulmonary function assessments were performed using centralized spirometry according to international standards. Baseline FEV1 was defined as the average of the pre-dose FEV1 measured at -45 minutes (min) and -15 min at day 1. A mixed model for repeated measures (MMRM), used for this analysis, included terms of treatment, baseline FEV1 measurements, smoking status at baseline, baseline inhaled corticosteroid (ICS) use, region, baseline FEV1 * visit interaction, and visit, treatment * visit interaction.
Time Frame: BL, Day 1: 5min, 15min, 1h, 2h, 4h, 6h, 8h, 11h55 min; Day 2: 23h15min, 23h45min; Day 15: -45min, -15min, 1h; Day 29: -45 min, -15min, 1h; Day 57: -45min, -15min, 1h; day 85: -45min, -15min, 5min, 15min, 1h, 2h, 4h, 6h, 8h, 11h; day 86: 23h15min; 23h45min
Population: Full Analysis Set (FAS): The FAS included all randomized participants who received at least one dose of study medication. Participants, who has both baseline and post baseline values for a given time point, were included in the analysis for that time point.
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | QVA149 | QAB149 | NVA237 | Placebo
Number analyzed (Participants) | 250 | 251 | 250 | 247
Liters
  day 1, 5 min (n=248,249,249,243) | 0.117 (0.0061) | 0.076 (0.0060) | 0.072 (0.0061) | -0.001 (0.0062)
  day 1, 15 min (n=248,251,249,244) | 0.160 (0.0070) | 0.090 (0.0069) | 0.126 (0.0070) | 0.005 (0.0070)
  day 1, 1 h (n=249,251,249,246) | 0.199 (0.0082) | 0.089 (0.0082) | 0.176 (0.0083) | 0.008 (0.0083)
  day 1, 2 h (n=249,249,248,246) | 0.237 (0.0091) | 0.109 (0.0091) | 0.197 (0.0092) | 0.030 (0.0092)
  day 1, 4 h (n=247,247,248,237) | 0.220 (0.0099) | 0.108 (0.0099) | 0.167 (0.0099) | 0.019 (0.0101)
  day 1, 6 h (n=247,246,244,239) | 0.181 (0.0103) | 0.085 (0.0104) | 0.135 (0.0104) | -0.005 (0.0106)
  day 1, 8 h (n=248,247,245,242) | 0.165 (0.0102) | 0.077 (0.0101) | 0.112 (0.0103) | -0.019 (0.0104)
  day 1, 11 h 55 min(n=242,243,244,239) | 0.116 (0.0114) | 0.029 (0.0114) | 0.066 (0.0114) | -0.045 (0.0115)
  day 2, 23 h 15 min (n=241,246,245,241) | 0.201 (0.0111) | 0.105 (0.0110) | 0.128 (0.0111) | 0.002 (0.0111)
  day 2, 23 h 45 min (n= 246,251,248,244) | 0.216 (0.0111) | 0.118 (0.0109) | 0.137 (0.0111) | 0.018 (0.0111)
  day 15, - 45 min (243,249,246,240) | 0.208 (0.0126) | 0.114 (0.0124) | 0.108 (0.0126) | -0.045 (0.0127)
  day 15, -15 min (n=243,248,246,241) | 0.238 (0.0124) | 0.143 (0.0123) | 0.132 (0.0124) | -0.025 (0.0124)
  day 15, 1 h (n=249,251,249,246) | 0.321 (0.0134) | 0.179 (0.0133) | 0.212 (0.0134) | -0.019 (0.0135)
  day 29, -45 min (n=243,249,246,240) | 0.213 (0.0132) | 0.127 (0.0131) | 0.117 (0.0132) | -0.030 (0.0133)
  day 29, -15 min (n=243,248,246,241) | 0.235 (0.0132) | 0.147 (0.0131) | 0.138 (0.0132) | -0.013 (0.0134)
  day 29, 1 h (n=249,251,249,246) | 0.320 (0.0135) | 0.170 (0.0135) | 0.216 (0.0136) | -0.004 (0.0137)
  day 57, -45 min (n=243,249,246,240) | 0.203 (0.0136) | 0.104 (0.0136) | 0.117 (0.0137) | -0.037 (0.0140)
  day 57, -15 min (n=243,248,246,241) | 0.224 (0.0136) | 0.125 (0.0135) | 0.147 (0.0136) | -0.014 (0.0139)
  day 57, 1 h (n=249,251,249,246) | 0.319 (0.0143) | 0.163 (0.0143) | 0.221 (0.0144) | -0.016 (0.0146)
  day 85, -45 min (n=243,249,246,240) | 0.187 (0.0134) | 0.090 (0.0135) | 0.096 (0.0135) | -0.032 (0.0138)
  day 85, - 15 min (n=243,248,246,241) | 0.199 (0.0138) | 0.109 (0.0137) | 0.123 (0.0138) | -0.018 (0.0141)
  day 85, 5 min (n=248,249,249,243) | 0.246 (0.0142) | 0.151 (0.0143) | 0.143 (0.0142) | -0.020 (0.0144)
  day 85, 15 min (n=248,251,249,244) | 0.269 (0.0141) | 0.153 (0.0142) | 0.179 (0.0141) | -0.001 (0.0145)
  day 85, 1 h (n=249,251,249,246) | 0.293 (0.0144) | 0.141 (0.0144) | 0.208 (0.0144) | -0.018 (0.0147)
  day 85, 2 h (n=249,249,248,246) | 0.315 (0.0146) | 0.159 (0.0147) | 0.216 (0.0148) | -0.001 (0.0150)
  day 85, 4 h (n=247,247,248,237) | 0.260 (0.0150) | 0.145 (0.0151) | 0.172 (0.0151) | -0.004 (0.0157)
  day 85, 6 h (n=247,246,244,239) | 0.226 (0.0149) | 0.122 (0.0150) | 0.139 (0.0151) | -0.011 (0.0155)
  day 85, 8 h (n=248,247,245,242) | 0.198 (0.0146) | 0.107 (0.0147) | 0.133 (0.0149) | -0.039 (0.0153)
  day 85, 11 h 55 min(n=242,243,244,239) | 0.163 (0.0147) | 0.078 (0.0150) | 0.105 (0.0150) | -0.073 (0.0154)
  day 86, 23 h 15 min (n=241,246,245,241) | 0.206 (0.0148) | 0.130 (0.0147) | 0.117 (0.0149) | -0.023 (0.0150)
  day 86, 23 h 45 min (n=246,251,248,244) | 0.221 (0.0144) | 0.144 (0.0144) | 0.132 (0.0146) | -0.012 (0.0149)

7. Secondary Outcome: Change From Baseline in FVC
Description: Pulmonary function assessments were performed using centralized spirometry according to international standards. Baseline FVC was defined as the average of the pre-dose FVC measured at -45 minutes (min) and -15 min at day 1. A mixed model for repeated measures (MMRM), used for this analysis, included terms of treatment, baseline FVC measurements, smoking status at baseline, baseline inhaled corticosteroid (ICS) use, region, baseline FEV1 * visit interaction, and visit, treatment * visit interaction.
Time Frame: as for outcome 6
Population: as for outcome 6
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | QVA149 | QAB149 | NVA237 | Placebo
Number analyzed (Participants) | 250 | 251 | 250 | 247
Liters
  day 1, 5 min (n=248,249,249,243) | 0.245 (0.0138) | 0.175 (0.0136) | 0.158 (0.0137) | -0.006 (0.0140)
  day 1, 15 min (n=248,251,249,244) | 0.318 (0.0154) | 0.185 (0.0153) | 0.238 (0.0155) | 0.009 (0.0155)
  day 1, 1 h (n=249,251,249,246) | 0.355 (0.0165) | 0.153 (0.0164) | 0.309 (0.0166) | 0.013 (0.0166)
  day 1, 2 h (n=249,249,248,246) | 0.395 (0.0181) | 0.214 (0.0180) | 0.324 (0.0182) | 0.044 (0.0183)
  day 1, 4 h (n=247,247,248,237) | 0.364 (0.0187) | 0.189 (0.0187) | 0.271 (0.0188) | 0.026 (0.0192)
  day 1, 6 h (n=247,246,244,239) | 0.316 (0.0186) | 0.159 (0.0188) | 0.244 (0.0189) | 0.004 (0.0192)
  day 1, 8 h (n=248,247,245,242) | 0.285 (0.0179) | 0.154 (0.0178) | 0.212 (0.0182) | -0.021 (0.0183)
  day 1, 11 h 55 min (n=242,243,244,239) | 0.235 (0.0188) | 0.093 (0.0188) | 0.125 (0.0188) | -0.060 (0.0190)
  day 2, 23 h 15 min (n=241,246,245,241) | 0.343 (0.0193) | 0.191 (0.0191) | 0.217 (0.0194) | 0.001 (0.0194)
  day 2, 23 h 45 min (n=246,251,248,244) | 0.355 (0.0195) | 0.196 (0.0192) | 0.229 (0.0194) | 0.027 (0.0195)
  day 15, -45 min (n=243,249,246,240) | 0.313 (0.0205) | 0.163 (0.0201) | 0.168 (0.0204) | -0.047 (0.0206)
  day 15, -15 min (n=243,248,246,241) | 0.358 (0.0207) | 0.201 (0.0204) | 0.198 (0.0207) | -0.020 (0.0207)
  day 15, 1 h (n=249,251,249,246) | 0.473 (0.0025) | 0.269 (0.0223) | 0.311 (0.0225) | -0.009 (0.0227)
  day 29, -45 min (n=243,249,246,240) | 0.320 (0.0217) | 0.194 (0.0216) | 0.188 (0.0217) | -0.025 (0.0220)
  day 29, -15 min (n=243,248,246,241) | 0.332 (0.0216) | 0.218 (0.0215) | 0.197 (0.0216) | -0.004 (0.0219)
  day 29, 1 h (n=249,251,249,246) | 0.449 (0.0224) | 0.259 (0.0223) | 0.322 (0.0225) | 0.008 (0.0227)
  day 57, -45 min (n=243,249,246,240) | 0.293 (0.0215) | 0.142 (0.0215) | 0.173 (0.0217) | -0.034 (0.0221)
  day 57, -15 min (n=243,248,246,241) | 0.298 (0.0223) | 0.167 (0.0222) | 0.222 (0.0224) | -0.009 (0.0229)
  day 57, 1 h (n=249,251,249,246) | 0.445 (0.0233) | 0.227 (0.0233) | 0.326 (0.0234) | -0.011 (0.0238)
  day 85, -45 min (n=243,249,246,240) | 0.252 (0.0223) | 0.121 (0.0224) | 0.143 (0.0225) | -0.029 (0.0229)
  day 85, -15 min (n=243,248,246,241) | 0.263 (0.0224) | 0.142 (0.0223) | 0.180 (0.0225) | -0.031 (0.0229)
  day 85, 5 min (n=248,249,249,243) | 0.331 (0.0243) | 0.215 (0.0244) | 0.225 (0.0243) | -0.048 (0.0247)
  day 85, 15 min (n=248,251,249,244) | 0.377 (0.0242) | 0.223 (0.0243) | 0.276 (0.0243) | -0.004 (0.0248)
  day 85, 1 h (n=249,251,249,246) | 0.400 (0.0243) | 0.209 (0.0243) | 0.295 (0.0244) | -0.023 (0.0248)
  day 85, 2h (n=249,249,248,246) | 0.414 (0.0244) | 0.218 (0.0245) | 0.301 (0.0247) | -0.001 (0.0251)
  day 85, 4 h (n=247,247,248,237) | 0.338 (0.0247) | 0.203 (0.0249) | 0.261 (0.0250) | 0.002 (0.0259)
  day 85, 6 h (n=247,246,244,239) | 0.305 (0.0239) | 0.164 (0.0240) | 0.211 (0.0241) | -0.011 (0.0248)
  day 85, 8 h (n=248,247,245,242) | 0.273 (0.0233) | 0.152 (0.0235) | 0.213 (0.0237) | -0.038 (0.0244)
  day 85, 11 55 min (n=242,243,244,239) | 0.233 (0.0239) | 0.131 (0.0243) | 0.197 (0.0243) | -0.093 (0.0250)
  day 86, 23 h 15 min (n=241,246,245,241) | 0.278 (0.0248) | 0.172 (0.0247) | 0.176 (0.0250) | -0.021 (0.0251)
  day 86, 23 h 45 min (n=246,251,248,244) | 0.298 (0.0240) | 0.199 (0.0239) | 0.210 (0.0244) | -0.017 (0.0248)

8. Secondary Outcome: Secondary: Change From Baseline in Standardized FEV1 AUC (0-4 h), FEV1 AUC (4-8h), FEV1 AUC (8-12h) and FEV1 AUC (0-12 h)
Description: Pulmonary function assessments were performed using centralized spirometry according to international standards. Baseline FEV1 was defined as the average of the pre-dose FEV1 measured at -45 minutes (min) and -15 min at day 1. A mixed model for repeated measures (MMRM), used for this analysis, included terms of treatment, baseline FEV1 measurements, smoking status at baseline, baseline inhaled corticosteroid (ICS) use, region, baseline FEV1 * visit interaction, and visit, treatment * visit interaction. The trapezoidal rule was used to calculate FEV1 AUC and then normalized to the length of time.
Time Frame: BL, day 1, 12 weeks
Population: Full Analysis Set: The FAS included all randomized participants who received at least one dose of study treatment. Participants, who had both baseline and post baseline values for a given time point, were included in the analysis for that time point.
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | QVA149 | QAB149 | NVA237 | Placebo
Number analyzed (Participants) | 250 | 251 | 250 | 247
Liters
  Day 1, AUC 0-4h (n=249,251,250,246) | 0.213 (0.0077) | 0.101 (0.0077) | 0.174 (0.0077) | 0.019 (0.0078)
  Day 1, AUC 4-8h (n=248,248,250,243) | 0.187 (0.0093) | 0.090 (0.0093) | 0.134 (0.0093) | -0.003 (0.0095)
  Day 1, AUC 8-12h (n=248,249,249,245) | 0.143 (0.0099) | 0.054 (0.0099) | 0.092 (0.0100) | -0.031 (0.0101)
  Day 1, AUC 0-12h (n=249,251,250,246) | 0.184 (0.0084) | 0.080 (0.0084) | 0.135 (0.0084) | -0.003 (0.0085)
  Week 12, AUC 0-4h (n=249,251,250,246) | 0.289 (0.0138) | 0.147 (0.0138) | 0.196 (0.0138) | -0.008 (0.0141)
  Week 12, AUC 4-8h (n=248,248,250,243) | 0.229 (0.0140) | 0.120 (0.0141) | 0.148 (0.0141) | -0.021 (0.0145)
  Week 12, AUC 8-12h (n=248,249,249,245) | 0.182 (0.0141) | 0.095 (0.0142) | 0.123 (0.0143) | -0.055 (0.0146)
  Week 12, AUC 0-12h (n=249,251,250,246) | 0.234 (0.0134) | 0.122 (0.0134) | 0.155 (0.0134) | -0.028 (0.0137)

9. Secondary Outcome: Transitional Dyspnea Index (TDI) Focal Score
Description: The Baseline Dyspnea Index (BDI) / TDI is an instrument used to assess a participant's level of dyspnea. The BDI and TDI each have three domains: functional impairment, magnitude of task and magnitude of effort. BDI domains were rated from 0 (severe) to 4 (unimpaired) and rates summed for baseline focal score ranged from 0 to 12; lower scores mean worse severity. TDI domains were rated from -3 (major deterioration) to 3 (major improvement) and rates summed for transition focal score ranged from -9 to 9; negative scores indicate deterioration. A TDI focal score of ≥1 was defined as a clinically important improvement from baseline.
Time Frame: BL, 12 weeks
Population: Full Analysis Set (FAS) The FAS included all randomized participants who received at least one dose of study treatment. Participants, who had both baseline and week 12 scores, were included in the analysis.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | QVA149 | QAB149 | NVA237 | Placebo
Number analyzed (Participants) | 233 | 238 | 232 | 222
score on a scale | 2.88 (0.251) | 1.98 (0.252) | 1.88 (0.252) | 0.85 (0.256)

10. Secondary Outcome: Secondary: Change From Baseline in Mean Daily Number of Puffs of Rescue Medication
Description: Participants completed an electronic diary (eDiary) twice daily at the same time in the morning and evening to record the number of puffs of rescue medication taken in the previous 12 hours. A negative change from baseline indicates improvement.
Time Frame: BL, 12 weeks
Population: Full Analysis Set (FAS) The FAS included all randomized participants who received at least one dose of study treatment. Participants, who had both baseline and week 12 values, were included in the analysis.
Measure: Least Squares Mean (Standard Error); unit: number of puffs
Arm/Group | QVA149 | QAB149 | NVA237 | Placebo
Number analyzed (Participants) | 243 | 242 | 242 | 235
number of puffs | -2.19 (0.150) | -2.05 (0.150) | -1.78 (0.151) | -1.04 (0.153)

11. Secondary Outcome: Secondary: Change From Baseline in Mean Total Daily Symptom Score, Mean Daytime Total Symptom Score and Mean Nighttime Total Symptom Score
Description: The participant recorded symptom scores twice daily in the eDiary. The daily clinical symptoms included: cough, wheezing, shortness of breath, sputum volume, sputum color, and night time awakening. The range of scores for each assessment is 0 to 3 where 0 indications No symptom and 3 indicates a Severe symptom. The maximum daytime total score is 27 and the maximum nighttime total score is 27. The total daily symptom score is obtained by adding the scores for the morning and evening symptoms for each day. The maximum possible total daily score is 54. A negative change from baseline indicated improvement.
Time Frame: BL, 12 weeks
Population: as for outcome 10
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | QVA149 | QAB149 | NVA237 | Placebo
Number analyzed (Participants) | 250 | 251 | 250 | 247
score on a scale
  total daily (n=243,242,242,235) | -1.34 (0.108) | -1.22 (0.108) | -1.09 (0.108) | -0.61 (0.110)
  total daytime (n=242,239,240,234) | -1.16 (0.105) | -1.05 (0.105) | -0.96 (0.105) | -0.53 (0.106)
  total nighttime (n=243,239,238,234) | -1.09 (0.107) | -1.01 (0.107) | -0.90 (0.108) | -0.41 (0.109)

ADVERSE EVENTS:
Arm/Group | QVA149 | QAB149 | NVA237 | Placebo
Serious Adverse Events (participants affected / at risk) | 6/250 | 5/251 | 12/251 | 13/248
Other Adverse Events (participants affected / at risk) | 60/250 | 51/251 | 62/251 | 71/248
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | QVA149 (N=250) | QAB149 (N=251) | NVA237 (N=251) | Placebo (N=248)
ANAEMIA (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
ANGINA PECTORIS (Cardiac disorders) | 0 | 1 | 0 | 0
CARDIAC FAILURE (Cardiac disorders) | 0 | 0 | 0 | 1
CARDIO-RESPIRATORY ARREST (Cardiac disorders) | 0 | 0 | 1 | 0
CARDIOPULMONARY FAILURE (Cardiac disorders) | 0 | 0 | 1 | 0
MYOCARDIAL INFARCTION (Cardiac disorders) | 1 | 0 | 0 | 0
INGUINAL HERNIA (Gastrointestinal disorders) | 0 | 0 | 1 | 0
PNEUMOPERITONEUM (Gastrointestinal disorders) | 0 | 0 | 1 | 0
CHEST PAIN (General disorders) | 1 | 0 | 0 | 0
OEDEMA PERIPHERAL (General disorders) | 0 | 0 | 1 | 0
HEPATIC FUNCTION ABNORMAL (Hepatobiliary disorders) | 0 | 1 | 0 | 0
EPIGLOTTITIS (Infections and infestations) | 0 | 0 | 1 | 0
LOWER RESPIRATORY TRACT INFECTION (Infections and infestations) | 0 | 1 | 0 | 0
PERIRECTAL ABSCESS (Infections and infestations) | 0 | 0 | 1 | 0
PNEUMONIA (Infections and infestations) | 1 | 0 | 0 | 0
SINUSITIS (Infections and infestations) | 0 | 0 | 0 | 1
UPPER RESPIRATORY TRACT INFECTION BACTERIAL (Infections and infestations) | 0 | 0 | 1 | 0
FEMUR FRACTURE (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1
GUN SHOT WOUND (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
HEPATIC ENZYME INCREASED (Investigations) | 0 | 0 | 0 | 1
DEHYDRATION (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
OSTEOARTHRITIS (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
BASAL CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
HEPATIC CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
METASTATIC MALIGNANT MELANOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
NON-SMALL CELL LUNG CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
PROSTATE CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
SQUAMOUS CELL CARCINOMA OF SKIN (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
CHRONIC OBSTRUCTIVE PULMONARY DISEASE (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 5 | 7
HAEMOPTYSIS (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
LUNG INFILTRATION (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
ERYTHEMA (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
HYPERTENSIVE CRISIS (Vascular disorders) | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | QVA149 (N=250) | QAB149 (N=251) | NVA237 (N=251) | Placebo (N=248)
ATRIAL FIBRILLATION (Cardiac disorders) | 3 | 0 | 0 | 0
CONSTIPATION (Gastrointestinal disorders) | 0 | 0 | 3 | 1
DIARRHOEA (Gastrointestinal disorders) | 0 | 1 | 3 | 0
DRY MOUTH (Gastrointestinal disorders) | 2 | 1 | 0 | 3
NAUSEA (Gastrointestinal disorders) | 0 | 1 | 2 | 4
SEASONAL ALLERGY (Immune system disorders) | 3 | 0 | 1 | 0
BRONCHITIS (Infections and infestations) | 3 | 5 | 5 | 3
INFLUENZA (Infections and infestations) | 2 | 4 | 1 | 1
NASOPHARYNGITIS (Infections and infestations) | 4 | 5 | 7 | 3
PHARYNGITIS (Infections and infestations) | 3 | 1 | 1 | 0
SINUSITIS (Infections and infestations) | 0 | 3 | 2 | 2
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 6 | 3 | 9 | 7
UPPER RESPIRATORY TRACT INFECTION BACTERIAL (Infections and infestations) | 3 | 6 | 2 | 6
URINARY TRACT INFECTION (Infections and infestations) | 3 | 0 | 4 | 2
VIRAL UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 4 | 2 | 3 | 5
CONTUSION (Injury, poisoning and procedural complications) | 2 | 3 | 1 | 1
BACK PAIN (Musculoskeletal and connective tissue disorders) | 4 | 2 | 1 | 2
MUSCULOSKELETAL CHEST PAIN (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 3
DIZZINESS (Nervous system disorders) | 0 | 0 | 3 | 0
HEADACHE (Nervous system disorders) | 1 | 5 | 2 | 4
INSOMNIA (Psychiatric disorders) | 3 | 1 | 1 | 0
CHRONIC OBSTRUCTIVE PULMONARY DISEASE (Respiratory, thoracic and mediastinal disorders) | 28 | 23 | 23 | 36
COUGH (Respiratory, thoracic and mediastinal disorders) | 3 | 3 | 1 | 6
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 3
OROPHARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 5 | 0 | 4 | 3
SPUTUM INCREASED (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 3
HYPERTENSION (Vascular disorders) | 3 | 2 | 3 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial or disclosure of trial results in their entirety.